CLINICAL TRIAL: NCT05120934
Title: A Randomized, Double-blind, Placebo Controlled, Dose Escalation Pilot Study Evaluating the Efficacy of Two Doses of Duloxetine and Amitriptyline in Interstitial Lung Disease-related Cough
Brief Title: Efficacy of Two Doses of Duloxetine & Amitriptyline in Interstitial Lung Disease-related Cough
Acronym: MACS-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vivek N Iyer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-009475
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Lung Disease
Keywords: ILD; cough; chronic cough; refractory; antitussives; IPF; fibrosis; UIP; NSIP; pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Cough; Chronic Cough; Fibrosis; Pulmonary Fibrosis | interventions — Amitriptyline; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the initial 8- week period, this will be a double-blind study. Both subjects and all study personnel (except for the research pharmacist) will be blind to the treatment assignment. Unblinding for both subjects and study investigators will occur at the end of the 8-week blinded treatment period.
  The subjects and all personnel involved with the conduct and the interpretation of the study, including the Investigators and other study personnel (except the research pharmacist) will be blinded to the treatment codes. Randomization data will be kept strictly confidential by the study statistician, and accessible only to authorized persons until the time of unblinding.
  Only in the case of an emergency, when knowledge of the investigational product is essential for the welfare of a subject, the principal investigator may unblind a subject's treatment assignment during the 8-week blinded treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Duloxetine and Placebo (Experimental): Subjects will receive 30mg of Duloxetine for blinded period 1 (first 4 week treatment period) and 30mg of Duloxetine plus 30mg Placebo for blinded period 2 (additional 4 weeks treatment period). After this, subjects will be unblinded and receive routine clinical care for follow up phase (up to 52 weeks).
  Interventions: Drug: Duloxetine 30 MG; Drug: Placebo 30 MG
- Duloxetine dose escalation (Experimental): Subjects will receive 30mg of Duloxetine for blinded period 1 (first 4 week treatment period) and 60mg of Duloxetine for blinded period 2 (additional 4 weeks treatment period). After this, subjects will be unblinded and receive routine clinical care for follow up phase (up to 52 weeks).
  Interventions: Drug: Duloxetine 30 MG; Drug: Duloxetine 60 MG
- Amitriptyline and Placebo (Experimental): Subjects will receive 25mg of Amitriptyline for blinded period 1 (first 4 week treatment period) and 25mg of Amitriptyline plus 30mg Placebo for blinded period 2 (additional 4 weeks treatment period). After this, subjects will be unblinded and receive routine clinical care for follow up phase (up to 52 weeks).
  Interventions: Drug: Amitriptyline 25 MG; Drug: Placebo 30 MG
- Amitriptyline dose escalation (Experimental): Subjects will receive 25mg of Amitriptyline for blinded period 1 (first 4 week treatment period) and 50mg of Amitriptyline for blinded period 2 (additional 4 weeks treatment period). After this, subjects will be unblinded and receive routine clinical care for follow up phase (up to 52 weeks).
  Interventions: Drug: Amitriptyline 25 MG; Drug: Amitriptyline 50 MG
- Placebo (Placebo Comparator): Subjects will receive 30mg of Placebo for blinded period 1 (first 4 week treatment period) and 60mg of Placebo for blinded period 2 (additional 4 weeks treatment period). After this, subjects will be unblinded and receive routine clinical care for follow up phase (up to 52 weeks).
  Interventions: Drug: Placebo 30 MG; Drug: Placebo 60 MG

INTERVENTIONS:
Drug: Amitriptyline 25 MG — 25 mg orally for 4 weeks
  Arms: Amitriptyline and Placebo; Amitriptyline dose escalation
Drug: Amitriptyline 50 MG — 50 mg orally for 4 weeks
  Arms: Amitriptyline dose escalation
Drug: Duloxetine 30 MG — 30mg orally for 4 weeks
  Arms: Duloxetine and Placebo; Duloxetine dose escalation
Drug: Duloxetine 60 MG — 60mg orally for 4 weeks
  Arms: Duloxetine dose escalation
Drug: Placebo 30 MG — 30mg tablet with no active study ingredient for 4 weeks
  Arms: Amitriptyline and Placebo; Duloxetine and Placebo; Placebo
Drug: Placebo 60 MG — 60mg tablet with no active study ingredient for 4 weeks
  Arms: Placebo

SUMMARY:
This research study is evaluating the effectiveness of escalating doses of Amitriptyline and Duloxetine in reducing cough frequency in patients with interstitial lung disease (ILD)-related cough.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-arm, dose escalation study of Duloxetine & Amitriptyline in subjects with interstitial lung disease-related chronic cough. Subjects will be screened during a period of up to 2 week and will undergo screening/ baseline cough monitoring. A total of 25 subjects who meet entry criteria will be randomly assigned in a 1: 1: 1: 1: 1 ratio to one of five treatment arms using stratified randomization in blocks of 5. Each arm will have two successive 4-week treatment periods (Blinded Period 1 & 2). After this, patients will be unblinded and receive routine clinical care. During the unblinded (routine clinical care) follow up phase; subjects will be initially offered the option of continuing amitriptyline or duloxetine based on their initial randomization arm. Subjects could also choose an alternative chronic cough therapy (e.g. pregabalin, gabapentin, 1% tetracaine lollipop or nebulized lidocaine or combination therapy).

Subjects in treatment arm 5, who received placebo during the 8 weeks blinded period will have a discussion regarding all available cough therapies. Patients will be offered the flexibility of therapy options during the unblinded follow up as they would during routine clinical care. Participation in the unblinded follow-up period will be optional.

Treatment Arm 1:

Blinded Period 1 (1st 4 weeks): 30mg of Duloxetine Blinded Period 2 (2nd 4 weeks): 30mg of Duloxetine & 30mg of Placebo Unblinded (routine clinical care) follow up period: (up to 52 weeks): Subjects will be offered routine clinical care management for their chronic cough

Treatment Arm 2:

Blinded Period 1 (1st 4 weeks): 30mg of Duloxetine Blinded Period 2 (2nd 4 weeks): 60mg of Duloxetine (2 pills of 30mg each) Unblinded (routine clinical care) follow up period: (up to 52 weeks): Subjects will be offered routine clinical care management for their chronic cough

Treatment Arm 3:

Blinded Period 1 (1st 4 weeks): 25mg of Amitriptyline Blinded Period 2 (2nd 4 weeks): 25mg of Amitriptyline + 25mg of Placebo Unblinded (routine clinical care) follow up period: (up to 52 weeks): Subjects will be offered routine clinical care management for their chronic cough

Treatment Arm 4:

Blinded Period 1 (1st 4 weeks): 25mg of Amitriptyline Blinded Period 2 (2nd 4 weeks): 50mg of Amitriptyline (2 pills of 25mg each) Unblinded (routine clinical care) follow up period: (up to 52 weeks): Subjects will be offered routine clinical care management for their chronic cough

Treatment Arm 5:

Blinded Period 1 (1st 4 weeks): 30mg of Placebo Blinded Period 2 (2nd 4 weeks): 60mg of Placebo (2 pills of 30mg each) Unblinded (routine clinical care) follow up period: (up to 52 weeks): Subjects will be offered routine clinical care management for their chronic cough

ELIGIBILITY:
Inclusion Criteria

* Have a diagnosis of interstitial lung disease according to the American Thoracic Society Guidelines
* Have a chronic cough for at least 3 months prior to the screening visit
* Patients should be on a stable dose of ILD-directed therapies for 3 months prior to enrollment and will be allowed to continue their ILD-directed therapies. These include -but are not limited to- corticosteroids, immunosuppressing agents such as azathioprine and mycophenolate, as well as antifibrotic medications including nintedanib and pirfenidone. Additional corticosteroids and adjustment of ILD-directed therapy doses is permitted if deemed appropriate by the treating physician
* Have a score of ≥ 40mm on the Cough Severity VAS at Screening.
* Women of child-bearing potential must agree to use 2 forms of acceptable birth control and make no donation of eggs from Screening through the end of the 8-week study period. Acceptable birth control methods include established use of oral, injected, or implanted hormonal methods of contraception; intrauterine device (IUD) or intrauterine system (IUS); tubal ligation; or male sterilization. Double-barrier method (diaphragm for female subject and condom for male partner with spermicidal) satisfies the requirement for 2 forms of acceptable birth control. When concordant with the preferred lifestyle of the subject, true and complete abstinence (not periodic abstinence) is acceptable.
* Male subjects and their partners of child-bearing potential must use 2 methods of acceptable birth control, 1 of which must be a barrier method, and make no donation of sperm from Screening until 3 months after the last dose of study drug at the end of 8 weeks.
* Have provided written informed consent.
* Are willing and able to comply with all aspects of the protocol.

Exclusion Criteria

* Current smoker (cigarettes, e-cigarettes or marijuana) or former smokers who have smoked within the past 12 months.
* Former smokers with > 20 pack-year history of smoking
* Ongoing treatment with an ACE-inhibitor that is considered as the potential cause of a subject's cough or requiring treatment with an ACE-inhibitor during the study or within 12 weeks prior to the Screening/Baseline Visit (Day -14 to Day 0).
* History of upper or lower respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Screening/Baseline Visit (Day -14 to Day 0)
* History of opioid use specifically prescribed for chronic cough within 2 weeks of the Screening/Baseline Visit (Day -14 to Day 0). Use of opioids for other indications (for example, to treat pain) is permitted.
* History of baclofen use specifically prescribed for chronic cough within 2 weeks of the Screening/Baseline Visit (Day -14 to Day 0). Use of baclofen for other indications (for example, to treat spasticity) is permitted.
* Presence of an untreated or undertreated cause (other than ILD) for the patient's chronic cough (as determined by the treating/referring physician per ACCP guidelines). e.g. uncontrolled asthma, GERD or post-nasal drainage that could potentially explain the patient's chronic cough.
* Requiring concomitant therapy with prohibited medications (listed below).
* Treatment with any pharmaceutical or biological investigational therapy (excluding coronavirus disease of 2019 (COVID) vaccination and COVID related monoclonal antibody therapy)
* Participation in another clinical trial that does not allow co-enrollment within 4 weeks prior to the Screening/Baseline Visit (Day -14 to Day 0)
* Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3x the upper limit of normal (ULN) during screening.
* Serum creatinine < 30 mL/min, hemodialysis or peritoneal dialysis
* Advanced liver disease as defined by the presence of cirrhosis and/or signs of portal hypertension
* History of previous hypersensitivity or intolerance to Duloxetine & Amitriptyline (patients who have previously been on either amitriptyline or duloxetine for chronic cough or other reasons and have tolerated the medication will be offered participation regardless of previous response to therapy).
* Currently pregnant or breastfeeding female subject.
* Presence of any medical condition or disability that the investigators believe could interfere with the assessment of safety or efficacy in this trial or compromise the safety of the subject.
* Planned or anticipated major surgical procedure or other activity that would interfere with the subject's ability to comply with protocol-mandated assessments (e.g., extended travel) during the subject's participation in the study.
* Currently taking either another SSRI, SNRI or MAO inhibitor which the patient cannot safely discontinue at least 2 weeks prior to the screening period.

Therapies that are prohibited during the 8-week blinded phase of the study:

The following therapies are prohibited from 2 week prior to the Screening/Baseline Visit (Day -14 to Day 0) through the end of the 8-week blinded treatment period.

* Opioids (of any kind including tramadol & codeine) specifically prescribed for treatment of cough
* Dextromethorphan
* Guaifenesin
* Chlorpheniramine
* Benzonatate
* Trazodone
* Pregabalin or gabapentin prescribed for chronic cough
* 1% tetracaine lollipops prescribed for chronic cough
* 4% nebulized lidocaine solution prescribed for chronic cough
* Any SSRI (selective serotonin reuptake inhibitor) e.g. bupropion, citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine.
* Any SNRI (serotonin-norepinephrine reuptake inhibitor) e.g. venlafaxine, desvenlafaxine, milnacipran, levomilnacipran
* Any Tricyclic antidepressant e.g. doxepin, clomipramine, nortriptyline, imipramine, protriptyline, amoxapine, trimipramine
* Any MAO (Monoamine oxidase) inhibitor. e.g. phenelzine, selegiline, isocarboxacid or tranylcypromine
* Patients who were previously prescribed either amitriptyline or duloxetine for chronic cough will be eligible for the study as long as they had discontinued the medication at least 12 weeks prior to the Screening/Baseline Visit (Day -14 to Day 0).

The following therapies are prohibited from 4 week prior to the Screening/Baseline Visit (Day -14 to Day 0) through the end of the 8-week blinded treatment period.

• Investigational biologic or pharmaceutical therapies (excluding COVID vaccination and COVID related monoclonal antibody therapy)

The following therapies are prohibited from 12 week prior to the Screening/Baseline Visit (Day -14 to Day 0) through the end of the 8-week blinded treatment period.

• Treatment with an ACE-inhibitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in awake objective cough frequency (at 4 & 8 weeks) | 4 weeks, 8 weeks
  The primary objective is to evaluate awake cough frequency at 4 and 8 weeks using the Leicester Cough Monitor. The acoustic cough monitor recordings will be analyzed using the Leicester Cough Monitor program V2.3-MB. This will also be performed at months 4, 6, 9 & 12 for subjects who choose to continue with the optional unblinded continuation of the study after the initial 8 weeks.

SECONDARY OUTCOMES:
Change in 24-Hour cough frequency | 4 weeks, 8 weeks
  This will also be evaluated using using the Leicester Cough Monitor and recordings will be analyzed using the Leicester Cough Monitor program V2.3-MB. All recordings will be kept confidential on a secure encrypted device. This will also be performed at months 4, 6, 9 & 12 for subjects who choose to continue with the optional unblinded continuation of the study after the initial 8 weeks.
Change in Cough Severity Diary score | 4 weeks, 8 weeks
  Measured using self-reported Cough Severity Diary that patients will fill at baseline and on daily basis. Change in self-reported Cough Severity Diary score at 4 and 8 weeks will be evaluated.
  Patients will be asked a series of 6 questions including and will provide an answer using a 5-point Likert scale (never, rarely, sometimes, often, constantly). The following questions will be evaluated:
  In the past 24 hours, how often did you cough? In the past 24 hours, how often did you experience coughing fits? In the past 24 hours, how severe was your cough? In the past 24 hours, how often did you have an urge to cough? In the past 24 hours, how often could you control your cough? In the past 24 hours, how severe was your pain from coughing?
  This will also be performed at months 4, 6, 9 & 12 for subjects who choose to continue with the optional unblinded continuation of the study after the initial 8 weeks
Change from Baseline in Leicester Cough Questionnaire (LCQ-acute) individual domain and total scores | 4 weeks, 8 weeks
  The Leicester Cough Questionnaire (Acute) is a validated tool for the assessment of chronic cough. It evaluates physical, psychological and social domains and how they are impacted by chronic cough. The physical domain consists of 8 questions, the psychological domain consists of 7 questions, and the social domain consists of 4 questions. The domain score will be calculated as the total score from questions in the domain divided by the number of items in the domain (range 1-7). The total score is the sum of individual domain scores and ranges from 3-21. The individual domain as well as the total score will be reported on weeks 4 & 8. This will also be performed at months 4, 6, 9 & 12 for subjects who choose to continue with the optional unblinded continuation of the study after the initial 8 weeks.
Change in Cough Severity Visual Analogue Scale (VAS) | 4 weeks, 8 weeks
  Scored on a 100 mm visual analogue scale at Screening/ Baseline visit (Day -14 to Day 0), and on Days 28, and 56. This will also be performed at months 4, 6, 9 & 12 for subjects who choose to continue with the optional unblinded continuation of the study after the initial 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek N Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20527349